CLINICAL TRIAL: NCT04475003
Title: Health Literacy Among Caregivers of Children With IgE-mediated Allergy With Risk of Anaphylaxis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, dr. Jasmine Leus, Kinderarts, Algemeen Ziekenhuis Maria Middelares
Other Study IDs: MMS2020.017
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Health Literacy; Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Teaching — Teaching session about anaphylaxis

SUMMARY:
Research on health literacy among caregivers of children with IgE-mediated allergy at risk of anaphylaxis (life-threatening allergic reaction). Health literacy is a person's ability to understand health information so that they can maintain or improve their health and quality of life (of themself and children).

The aim of the study is to test the general knowledge of anaphylaxis. Furthermore we test the extent to which caregivers consider themselves able to recognize and to treat anaphylaxis.

ELIGIBILITY:
Inclusion Criteria:

* caregivers of children with IgE-mediated allergy with risk of anaphylaxis (adults, grandparents, school caregivers etc.).
* minimum 18 years old.
* signed informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For each child that is known with IgE-mediated allergy with risk of anaphylaxis parents can invitate 4 Caregivers of children with IgE-mediated allergy with risk of anaphylaxis (adults, grandparents, school caregivers etc.).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
General knowledge of anaphylaxis. | 1.5 year
  Knowledge Quiz

SECONDARY OUTCOMES:
The extent to which caregivers consider themselves able to recognize and to treat anaphylaxis. | 1.5 year
  Numeric scoring scale (0= cannot do at all, 5= highly certain can do)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine S Leus, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- Algemeen Ziekenhuis Maria Middelares, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No